CLINICAL TRIAL: NCT05476003
Title: Role of Bilateral Ultrasound Guided Superficial Cervical Plexus Block as a Part of Enhanced Recovery After Thyroid Surgery
Brief Title: Bilateral Ultrasound Guided Superficial Cervical Plexus Block After Thyroid Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Fatma Elsamahy, Dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 34751/6/21
Record Dates: First submitted 2022-07-24; First posted 2022-07-27 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Bilateral Ultrasound Guided Superficial Cervical Plexus Block; Thyroid Surgery; Enhanced Recovery
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All blocks will be performed by the same anesthesiologist while the measurements will be recorded by anesthesiologist who has no idea about patient allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Technique (Sham Comparator): Patients will receive general anesthesia plus Ultrasound-guided Bilateral superficial cervical plexus block with injection of 10 ml normal saline bilaterally.
  Interventions: Procedure: Ultrasound-guided Bilateral superficial cervical plexus block; Drug: Midazolam
- Ultrasound-guided Bilateral superficial cervical plexus block (Active Comparator): Patients will receive general anesthesia plus Ultrasound-guided Bilateral superficial cervical plexus block with injection of total volume 10 ml containing Bupivacaine 0.25% (5 ml Bupivacaine 0.5 % and 5 ml normal saline).
  Interventions: Procedure: Ultrasound-guided Bilateral superficial cervical plexus block; Drug: Midazolam

INTERVENTIONS:
Procedure: Ultrasound-guided Bilateral superficial cervical plexus block — This nerve block is typically performed in the supine or semi-sitting position, with the head turned slightly away from the side to be blocked to facilitate operator access.
  Under strict aseptic condition, the linear ultrasound transducer should be placed on the lateral neck, overlying the sternocleidomastoid muscle at the level of its midpoint (approximately the level of the cricoid cartilage). Once the sternocleidomastoid muscle has been identified, the transducer is moved posteriorly until the tapering posterior edge is positioned in the middle of the screen.
  Once the plexus has been identified and using In-Plane approach, the needle is passed from medial to lateral through the skin, platysma and investing layer of deep cervical fascia and the tip is placed adjacent to the plexus.
  Following negative aspiration, 1 mL of local anesthetic is injected to confirm the proper injection site. The remainder of the local anesthetic (5ml) is administered to envelop the plexus.
Drug: Midazolam — All patients will be premedicated with Midazolam (0.02mg/Kg).

SUMMARY:
Evaluating ultrasound guided Bilateral Superficial Cervical Plexus Block as a part of enhanced recovery after thyroid surgery using Quality of Recovery-15 scale as a method for assessment of quality of recovery.

DETAILED DESCRIPTION:
Surgery of the thyroid gland is increasingly popular performed as ambulatory procedures in many countries. Postoperative wound pain is a common complication, especially within 24 hr after thyroid surgery, which may delay discharge or even unplanned readmissions following day surgery.

Several strategies, including local and regional anesthesia, are now performed as core components of multimodal analgesia for postoperative pain. Adequate postoperative pain relief is imperative to improve functional outcome, accelerate early ambulation and discharge from the hospital.

Ultrasound-guided superficial cervical plexus block was introduced by Tran et al . The main advantages of Ultrasound-guided superficial cervical plexus block include: provide real-time visualization of anatomical structures, reduced volumes of local anesthetics, and avoid inadvertent damage or accidental puncture of vessels.

Owing to its feasibility and efficacy, ultrasound-guided Bilateral superficial cervical plexus block is a technique for providing adequate regional analgesia during thyroidectomy with improvement of patient recovery.

Quality of recovery after anesthesia is an important measure of the early postoperative health status of patients. Based on extensive clinical and research experience with the 40-item Quality of Recovery-40, the strongest psychometrically performing items from each of the five dimensions of the Quality of Recovery-40 were selected to create a short-form version. The Quality of Recovery-15 provides a valid, extensive, and yet efficient evaluation of postoperative Quality of Recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21 to 65 years
* American Society of Anesthesiologists physical status I or II.
* Scheduled for elective thyroid surgery.

Exclusion Criteria:

* Patient refusal to participate.
* Patients with history of allergy to local anesthetics.
* Patients with history of chronic use of pain killers .
* Patients presented with mental dysfunction.
* Patients with coagulation disorders.
* Patients presented with skin or soft tissue infection at the proposed site of needle Insertion.
* Patients with Chronic Obstructive Pulmonary Disease or Body Mass Index more than 40.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-08-15 (Estimated); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery | 24 hours postoperatively.
  Improvement of the quality of recovery assessed using the 15-item quality of recovery questionnaire. The Quality of Recovery-15 included 15 items 1-Breathing 2-Food 3-Rest 4-Sleep 5-Hygiene 6-Communication 7-Support 8-Return to work 9-Feeling comfortable and in control 10-Feeling of general well-being 10-Moderate pain 12-Severe pain 13-Nausea/Vomitting 14-Worry/Anxiety 15-Feeling sad or depressed .
  Each item will be assessed using a10-point numerical rating scale. The total score of Quality of Recovery-15 ranges from 0 (extremely poor recovery) to 150 (all excellent recovery).

SECONDARY OUTCOMES:
Postoperative analgesia | 24 hours postoperatively
  Postoperative analgesia defined by the visual analogue scale score 30 min after arrival to recovery room then after 2, 4, 6, 12, 24 hr. If visual analogue scale˃ 3 , morphine 3 mg will be given .
Opioid consumption | 24 hours postoperatively
  Total post operative opioid requirement will be recorded
Diaphragmatic Excursion | 24 hours postoperatively
  Diaphragmatic Excursion assessed by Ultrasound